CLINICAL TRIAL: NCT05438953
Title: Follow-up of People at Risk of Monkeypox Infection: a Prospective Cohort Study
Acronym: MonkeyVax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP220580; 2022-002352-39 (Other: ANSM)
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Monkey Pox; Monkey Diseases
Keywords: Monkeypox; Vaccines; Prevention; Post exposure vaccination (PEP); Pre exposure vaccination (PrEP)
MeSH Terms: conditions — Mpox, Monkeypox; Monkey Diseases | interventions — Vaccination; MVA vaccine; smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP Vaccinated (Experimental)
  Interventions: Biological: Vaccination with MVA vaccine ( IMVANEX® and JYNNEOS®)
- PrEP Vaccinated (Experimental)
  Interventions: Biological: Vaccination with MVA vaccine ( IMVANEX® and JYNNEOS®)

INTERVENTIONS:
Biological: Vaccination with MVA vaccine ( IMVANEX® and JYNNEOS®) — Participant of these arm will receive 2 doses of MVA vaccine spaced 28 days apart

SUMMARY:
Since one month (first case confirmed the 05/06/2022), some cases of non-imported were reported by Portuguese and British authorities then in several Europeans countries, the US and the Canada. The 05/19/2022, a first case of Monkeypox was confirmed in France. The 06/01/2022, "Santé Publique France" (SPF) declared 33 confirmed cases of Monkeypox without a direct interaction with people returning from endemic area. No deaths are currently recorded.

Currently, data on efficiency of modified vaccinia Ankara virus (MVA) used in post-exposure prophylaxis are few. The Centers for Disease Control and Prevention (CDC) consider that 2 doses of MVA vaccine used in post-exposure vaccination do not prevent totally the infection but consider that one rapid vaccination of high-risk contacts could reduce the severity of symptoms.

In order to clarify clinical impact and safety of PEV, it is proposed to set up a national cohort including people at risk of Monkeypox infectionfalling within the indications for vaccination, i.e. seen within 14 days of last contact for post-exposition (PEP) cases and also in prevention :pre-exposition ( PrEP)cases.

The purpose of this study is to estimate the failure rate of the vaccinationby the VMA vaccine in PEP or PrEP administration in people at risk of Monkeypox infection after one dose.

DETAILED DESCRIPTION:
Indication for Post-Exposure vaccination (PEP) :

PEP has demonstrated its interest in different situations, in particular rabies, tetanus or hepatitis B, as recalled in the report "Guide for post-exposure immunization: vaccination and immunoglobulin" of the High Committee for Public Health in 2016.

For Monkeypox, the PEV was used in 2018 and 2019 in UK, when several import cases were discovered. In 2018, 3 cases were diagnosed and 154 contact cases identified (including 147 healthcare professionals). In total, 131 people have accepted the PEV (including 126 healthcare professionals) and 1 single case among healthcare professionals, having been exposed for 6 to 7 days. In 2019, following an imported case, 17/18 contacts (including children) accepted EPV. No secondary cases or serious adverse effects have been reported.

Several countries have recommended EPV as part of Monkeypox.

Indication for Pre-Exposure vaccination (PrEP):

Since 2022/07/07, in addition to PEP vaccination, HAS recommends vaccination (PrEP) to people at very high risk of infection:

* Men who have sex with men (MSM) reporting multiple partners and trans people reporting multiple sexual partners
* People in prostitution
* Professionals in places of sexual consumption, regardless of the status of these places.

In France, the Haute Autorité de Santé (HAS) recommends that pre-exposure vaccination with 3rd generation MVA-BN vaccines (Imvanex and Jynneos) be offered to female partners who are occasional or who share the same living environment as people at very high risk of exposure, including MSM reporting multiple sexual partners and trans people reporting multiple sexual partners, people in a situation of prostitution and professionals in places of sexual consumption, regardless of the status of these places.

HAS also recommends the implementation of a reactive vaccine strategy with the 3rd generation vaccine administered in 2 doses spaced 28 days apart. For people who received smallpox vaccination with a 1st generation vaccine before 1980, only one dose of MVA vaccine should be administered. For immunocompromised subjects, regardless of their vaccination status, a three-dose schedule, each 28 days apart, is recommended. In post-exposure (PEP) the first dose being ideally administered within 4 days after the risky contact and at most 14 days after the risky contact.

Currently, data on the efficacy of the MVA vaccine used in post-exposure prophylaxis are few. The Centers for Disease Control and Prevention considers it unlikely that 2 doses of MVA vaccine used in PEV will completely prevent infection but believes that rapid vaccination of at-risk contacts could reduce the severity of symptoms.

In France, the definitions for identifying contact persons are :

1. Contact at risk:

   * Anyone who has had unprotected direct physical contact, i.e. without wearing surgical masks and FFP2, without using hygiaphones and vis-à-vis direct physical contact, without wearing waterproof gloves (latex, nitrile, rubber) with damaged skin or biological fluids of a probable or confirmed symptomatic case, whatever the circumstances, including acts of medical or paramedical care, or sharing of toilet utensils, or contact with textiles (clothing , bath linen, bedding) or dirty dishes used by the probable or confirmed symptomatic case.
   * Anyone who has had unprotected contact at less than 2 meters for 3 hours with a probable or confirmed symptomatic case (e.g. close or intimate friend, transport neighbour, office neighbour, people sharing the same living space with no intimate ties, act of care or hygiene, school and university environment, sports club, etc.). "
2. Confirmed case:

   * A positive qPCR or RT-PCR result specific for the MKPXV virus
   * A positive result in generic qPCR of the genus Orthopoxvirus, in a person presenting recent risks of exposure to the MKPXV virus in the 3 weeks preceding the onset of the signs (returning from a trip to an endemic zone or where the virus is circulating or at-risk contact of a person returning from a trip to an endemic zone or where the virus is circulating, contact person at risk of a probable or confirmed case).

In order to specify the clinical interest and the safety of MVA vaccination administered in PEP or PrEP in people at risk of infection, it is proposed to set up a national cohort including contact cases falling within the indications for vaccination, i.e. seen within 14 days after the last contact but also people vaccinated with PrEP representing the majority of vaccinations currently.

ELIGIBILITY:
Inclusion Criteria:

- PEP group : Be a contact at risk of exposure to the Monkeypox virus as recommended by the HAS within at less 14 days and not vaccinated OR Be a contact at risk of exposure to the Monkeypox virus as recommended by the HAS within at less 14 days and who received the first injection of PEV less than 28 days ago

- PrEP group : Be identified as belonging to the groups most exposed to MPXV, as defined by HAS, but not be a contact person at risk and not have received an MVA vaccine

- Signature of informed consent

Exclusion Criteria:

* Be under guardianship or curatorship
* No covered by social security
* Subject to a legal protection measure
* Have a contraindication to Monkeypox vaccination
* Have a known or suspected allergy to one of the components of the vaccine- Diagnosis of Monkeypox

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of failure of MVA vaccine | D28 after the first injection for PEP and between 14 days and 3 month for PrEP
  Positive PCR MKPXV

SECONDARY OUTCOMES:
Assess early vaccine humoral immunogenicity | Day 0, Day 7; Day 14 after the first injection (Day 0)
  Poxvirus antibody titer serological and neutralizing
Estimate the short-term vaccine failure rate after a risky contact | 28 days after the first injection
  Cumulative incidence of probable cases or confirmed cases within 28 days after the 1st dose of vaccine: among participants vaccinated in PEP
Estimate long-term vaccine failure rate (among PrEP or PEP participants) | up to 1 year after the first injection
  Cumulative incidence of probable cases or confirmed cases occurring at least 14 days and up to 1 year after the 1 redose of vaccine in participants vaccinated with PEP or PrEP
Evaluate the proportion of failures and their clinical presentations according to the time between exposure and vaccination | Day 0, Day 7, Day 14, Day 28, 1 month, Day 43 and 3 months
  Proportion of failure and clinical presentation in vaccinated group <4days after exposure, 4 to 14 days and >14 days
Effectiveness of MVA vaccination (PEP vs PrEP) | Day 0, Day 7; Day 14, Day 28, Month 1, 43 Days and 3 Months
  Comparison of the number of infections in PEP vaccinated versus PrEP
Effectiveness of MVAvaccination (PEP and PrEP) | D0, D7; D14, D28, Month 1, 43 Days et 3 Months
  Comparison of the number of infections in PEP and PrEP vaccinated and the number of infections in unvaccinated
Assess vaccine reactogenicity after each dose of vaccines | up to 1 year after the first injection of PEV
  Any adverse effects, local and systemic reactions occurring
Assess the acceptability of post-exposure vaccination | Day 0 (inclusion)
  Proportion of people accepting vaccination and reasons for non-acceptance
Prevalence of sexually transmitted infections | Day 0
  Seropositivity HIV, VHA (IgM), VHB (Ac-Hbs positive + Ac-Hbc positive), HCV, Syphilis
Assess the transmissibility of asymptomatic forms | D0, D7, D14, D28, D43 , M3, M6 and M12 after the first injection (D0)
  Detection of monkeypox virus in biological samples, Monkeypox PCR
Titre of antibodies directed against the Monkeypox virus | D7, D14, D28, D43 and M3 after the first injection (D0)
  Study the humoral immunogenicity of the vaccine and the factors associated with the humoral immune response
Cellular immunity to PEP and PrEP vaccination | D0, D10, M3 after the first injection (D0)
  Study of cellular immunity to MVA vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Liem binh LUONG NGUYEN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CIC Cochin-Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No